CLINICAL TRIAL: NCT02929043
Title: Psychophysical Characterization and Brain Correlates of Dentine Hypersensitivity
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: G1
Record Dates: First submitted 2016-01-08; First posted 2016-10-10 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dentine hypersensitivity subjects
  Interventions: Other: air puffs

INTERVENTIONS:
Other: air puffs

SUMMARY:
Up to date, devices capable of delivering controlled, calibrated, non-contact cold air stimuli in a MR environment are unavailable for quantitative sensory testing. This project therefore aimed at designing and constructing a novel MR-compatible, computer-controlled cold air stimulation device that produces air puffs in a broad flow and cold temperature range. By means of this device, detailed psychophysically testing and subsequent brain scanning of dentine hypersensitivity (DH) subjects will be possible to gain new insights about DH mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age and between 18 - 60

Exclusion Criteria:

* Caries
* Defective restorations
* Full crowns
* Orthodontic bands
* Bleeding on probing and periodontal pockets deeper than 3 mm
* Subjects with gross periodontal disease or treatment of periodontal disease in the past 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Dentine hypersensitivity (DH) is characterized by a short, sharp pain arising from exposed dentin.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Subjective ratings using the BORG scale | May 1, 2016
  individual subject perception ratings will be recorded by means of an adapted BORG scale. For reliability, intraclass correlations will be used covering 3-4 measures within a 3-4-weeks period.
blood oxygenation level dependent (BOLD) response | October 1, 2016
  Changes in blood oxygenation level (indirect measure of neural activity) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Ettlin, MD,DMD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Center of Dental Medicine, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes